CLINICAL TRIAL: NCT06255301
Title: Collection of Ocular Surface Impressions Cytology of the Living Eye From Patients With Dry Eyes or Limbal Stem Cell Deficiency.
Acronym: ESSO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Laboratoire Biologie, Ingénierie et Imagerie de la Greffe de Cornée (BiiGC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19CH218; 2020-A00139-30 (Other: ANSM)
Record Dates: First submitted 2024-02-02; First posted 2024-02-13 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Eye Diseases
Keywords: biomarkers; limbic stem cell deficiency; dry syndrome; EYEPRIM
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: 150 patients with eye diseases other than dry eye syndrome or limbal stem cell deficiency will be included.
  Interventions: Diagnostic Test: EYEPRIM
- dry eye syndrome: 100 patients with dry eye syndrome will be included.
  Interventions: Diagnostic Test: EYEPRIM
- limbal stem cell deficiency: 50 patients with limbal stem cell deficiency will be included.
  Interventions: Diagnostic Test: EYEPRIM

INTERVENTIONS:
Diagnostic Test: EYEPRIM — Collection of conjunctival impressions using the EC(European Conformity )-marked EYEPRIM device . This device enables cells to be collected the superficial ocular surface cells by applying a membrane for few seconds to the ocular surface.

SUMMARY:
In order to develop innovative biomarkers for the diagnosis of two ocular surface pathologies, Dry Syndrome (DS) and Limbic Stem Cell Deficiency (LSCD), human cells from the ocular surface will be collected in order to test these biomarkers ex vivo.

DETAILED DESCRIPTION:
To collect them, cytological fingerprints of the ocular surface are made using filter paper applied to the surface using a commercially available EC (European Conformity)-marked medical device, called EYEPRIM.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security scheme
* Age 18 years or older
* Presenting a Dry Syndrome, a limbic stem cell deficiency (clinical diagnosis) or another pathology (control).
* Signature of Consent

Exclusion Criteria:

* Major blepharospasm making examination impossible
* Pregnant women
* Breastfeeding women
* Protected Persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 50 patients with limbal stem cell deficiency
  * 100 patients with dry eye syndrome
  * 150 patients with eye diseases other than dry eye syndrome or limbal stem cell deficiency
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Ocular surface impression cytology collected from patients suffering from dry eye syndrome, limbal stem cell deficiency or other pathologies (control). | day one
  Collection of cells from the ocular surface by performing a cytological imprint of the ocular surface

CONTACTS AND LOCATIONS:
Overall Officials: Gilles THURET, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No